CLINICAL TRIAL: NCT02449785
Title: Assessment of Lung Involvement in Cystic Fibrosis Patients Using 1.5T MR Imaging With Ultrashort Echo Time (UTE) Pulse Sequences
Brief Title: Assessment of Cystic Fibrosis Lung Involvement With UTE Pulse Sequences
Acronym: MucoIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX2014/11
Record Dates: First submitted 2015-05-13; First posted 2015-05-20 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; MRI; UTE; CT; Exacerbation; Quality of life; Pulmonary function
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cystic fibrosis adults (Experimental)
  Interventions: Device: MR measurements of lung morphological changes in cystic fibrosis (Avanto dot, Siemens); Device: CT measurements of lung morphological changes in cystic fibrosis

INTERVENTIONS:
Device: MR measurements of lung morphological changes in cystic fibrosis (Avanto dot, Siemens)
Device: CT measurements of lung morphological changes in cystic fibrosis

SUMMARY:
Non-invasive assessment of lung involvement is a crucial issue for the follow-up of cystic fibrosis patients. Currently, CT is the method of reference to evaluate and quantify the lung morphological changes in cystic fibrosis adults but it remains a radiation-based technique. MRI with ultrashort echo time (UTE) pulse sequences is a promising non-ionizing alternative for lung imaging. The investigators' objective is to evaluate cystic fibrosis lung involvement using CT and MRI-UTE, and to test the agreement between both techniques.

DETAILED DESCRIPTION:
Cystic fibrosis is a recessive autosomic fatal disease, affecting about 6000 people in France. Thanks to progress in symptomatic care, median survival is increasing. The lung involvement is the most common and responsible for most deaths. The evaluation of respiratory disease severity is based on pulmonary functional tests (PFT) and imaging. Multi-slice computed tomography (CT) is the method of reference to quantify lung involvement in cystic fibrosis. It detects respiratory lung involvement earlier than PFT, and it reveals lesions associated with the onset of respiratory exacerbations, the mortality increase and the reduction of quality of life. However CT provides ionizing radiation, thus limiting the possibility of long-term follow-up. MRI is a non-ionizing 3D imaging technique; nevertheless, lung MRI is technically challenging with the result that it is currently not used in routine practice. Indeed, both low proton density and susceptibility effects lead to very low signal intensity derived from lung parenchyma. Recently, pulse sequences with ultrashort echo time (UTE) have been implemented by the use of half radio-frequency excitations and radial projection reconstruction. These UTE sequences make it theoretically possible to retrieve more signal from the lung parenchyma. The investigators aim at using 3D T1-weighted UTE pulse sequences on a 1.5T magnet (Avanto dot, Siemens) in cystic fibrosis patients in order to assess lung involvement severity. Thirty three cystic fibrosis adults are expected to take part in the study. All will benefit from PFT, CT and MRI. The investigators' strategy is to establish a semi quantitative score of pulmonary severity (Helbich score) using MRI and CT in subjects, testing for correlations between MRI and CT measurements and assessing the reproducibility of lung lesions quantification using MRI. The investigators' objective is to demonstrate that MRI-UTE pulse sequence at 1.5T is accurate and reproducible in evaluating and quantifying pulmonary involvement in cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis adults
* written informed consent

Exclusion Criteria:

* Subjects without any social security or health insurance
* Pregnancy
* MRI contraindications: Magnetically activated implanted devices (cardiac pacemakers, insulin pumps, neurostimulators, cochlear implants), metal inside the eye or the brain (aneurysm clip, ocular foreign body), cardiac valvular prosthesis (Starr-Edwards pre-6000), subject with claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Agreement between MRI and CT for scoring lung involvement in cystic fibrosis | During MRI and CT, Day one
  MRI and CT evaluation of lung lesions quantification in cystic fibrosis will be assessed by 2 blind radiologists.
  Agreement between both evaluation will be assessed during statistical analyses after study completion.

SECONDARY OUTCOMES:
Cystic fibrosis lesions scoring extracted from CT and MR images | During MRI and CT, Day one
  MRI and CT evaluation of lung lesions quantification in cystic fibrosis will be assessed by 2 blind radiologists.
  Agreement between both evaluation will be assessed during statistical analyses after study completion.
MRI cystic fibrosis reproductibility scoring over the time | During MRI, Day one
  MRI cystic fibrosis scoring will be assessed a second time the same blind radiologist
Correlation between MRI cystic fibrosis scoring and PFT indexes | Day one
Correlation between MRI cystic fibrosis scoring and exacerbation number | 12 month after Day one
Correlation between MRI cystic fibrosis scoring and quality of life | Day one and 12 month after Day one
Evolution of MRI cystic fibrosis scoring after one year | 12 month after Day one

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bordeaux, Pessac, France

REFERENCES:
- [Derived] Benlala I, Point S, Leung C, Berger P, Woods JC, Raherison C, Laurent F, Macey J, Dournes G. Volumetric quantification of lung MR signal intensities using ultrashort TE as an automated score in cystic fibrosis. Eur Radiol. 2020 Oct;30(10):5479-5488. doi: 10.1007/s00330-020-06910-w. Epub 2020 May 15. PMID 32415586